CLINICAL TRIAL: NCT00287859
Title: Phase I Study of Weekly Topotecan in Women With Progressive or Recurrent Ovarian Cancer and a Poor Performance Status
Brief Title: Topotecan in Treating Patients With Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to low accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Levi Downs, Jr, MD, Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS039; UMN-WCC-39 (Other: Women's Cancer Center, University of Minnesota)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: fallopian tube cancer; peritoneal cavity cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escalating Cohorts (Experimental): Patients receive topotecan intravenously (IV) over 30 minutes on days 1, 8, 15, 22, and 29. Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 6 patients will be treated at the MTD.
  Interventions: Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: topotecan hydrochloride — intravenously (IV) over 30 minutes on days 1, 8, 15, 22, and 29.
  Other Names: Hycamtin(R)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemotherapy drugs may have different effects in patients who have a poor performance status.

PURPOSE: This phase I trial is studying the side effects and best dose of topotecan in treating patients with progressive or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer with a poor performance status.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of weekly topotecan in patients with progressive or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer and a poor performance status.

Secondary

* Estimate the response rate of women with poor performance status for use in future clinical trials.

OUTLINE: This is a dose-escalation study.

Patients receive topotecan intravenously (IV) over 30 minutes on days 1, 8, 15, 22, and 29. Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 6 patients will be treated at the MTD.

Patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer

  * Progressive or recurrent disease
* Received ≥ 1 prior course of chemotherapy
* Measurable or evaluable disease OR disease assessable by CA 125, defined as CA 125 > normal that has increased over 2 readings > 14 days apart
* Karnofsky performance status 10-50%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 mg/dL
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* SGOT ≤ 3 times ULN
* Life expectancy ≥ 12 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use accepted and effective non-hormonal contraception

Exclusion Criteria:

* Other neoplasm within the past 5 years except for nonmetastatic, nonmelanoma skin cancers, carcinoma in situ of the cervix, or cancer cured by surgery or chemotherapy
* Septicemia, severe infection, or acute hepatitis
* Severe gastrointestinal bleeding, defined as requiring a blood transfusion or hospitalization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose

CONTACTS AND LOCATIONS:
Overall Officials: Levi S. Downs, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States